CLINICAL TRIAL: NCT06845163
Title: Clinical Study on the Efficacy of Oral Dapagliflozin Combined With Intravitreal Injection of Anti-Vascular Endothelial Growth Factor in Patients With Diabetic Macular Edema
Brief Title: Randomized Clinical Trial to Evaluate the Effect of Dapagliflozin in Patients With Diabetic Macular Edema
Acronym: DAPA-DME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0202071
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Macular Edema; Center-involved Diabetic Macular Edema
Keywords: Diabetic Macular Edema; center-involved diabetic macular edema; Anti-VEGF; Aflibercept; EYLEA; Dapagliflozin; Forxiga; SGLT2 inhibitor
MeSH Terms: interventions — dapagliflozin; aflibercept

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): The treatment group will receive oral dapagliflozin 10 mg daily in addition to standard of care intravitreal aflibercept injections.
  Interventions: Drug: Dapagliflozin; Drug: Anti-VEGF drug
- Control group (Active Comparator): The control group will receive standard of care intravitreal aflibercept injections.
  Interventions: Drug: Anti-VEGF drug

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg will be given orally once daily for three months.
  Other Names: Forxiga 10 mg
  Arms: Treatment group
Drug: Anti-VEGF drug — Aflibercept 2 mg (0.05 ml) will be administered by intravitreal injection every month for three consecutive months.
  Other Names: Aflibercept (Eylea)

SUMMARY:
The purpose of this clinical study is to explore the efficacy of dapagliflozin as an adjunct to intravitreal anti-vascular endothelial growth factor (anti-VEGF) for enhanced reduction of retinal thickness and vision improvement in patients with diabetic macular edema. The main question the study aims to answer is: Does dapagliflozin reduce the thickness of the macula when combined with the standard of care intravitreal anti-VEGF therapy more than the intravitreal anti-VEGF therapy alone?

DETAILED DESCRIPTION:
Some evidence in the literature suggests that sodium glucose co-transporter 2 (SGLT2) inhibitors may be beneficial in reducing diabetic macular edema. The objective of this clinical trial is to investigate the efficacy and safety of dapagliflozin when combined with intravitreal aflibercept injections in the management of patients with type II diabetes mellitus and center-involved diabetic macular edema (ci-DME). This randomized, double-blind, parallel group, active control design, clinical trial, is investigating the effect of oral dapagliflozin 10 mg given once daily in addition to intravitreal aflibercept versus intravitreal aflibercept alone on reducing macular central subfield thickness (CST) and improving visual acuity in diabetic patients with ci-DME.

ELIGIBILITY:
Inclusion criteria:

* Type II diabetes mellitus patients, treated with premixed insulin and metformin, and diagnosed with center-involved diabetic macular edema (CiDME)
* Presence of retinal thickening involving the center of the fovea (CiDME) in the study eye on Optical Coherence Tomography (OCT) Heidelberg Spectralis; If both eyes are eligible, the eye with the greater central subfield thickness on OCT is selected as the study eye.
* Decreased visual acuity primarily attributable to DME
* Clear ocular media and pupillary dilation for adequate retinal imaging
* Ability to understand the study procedures and willingness to provide written informed consent

Study participant exclusion criteria:

* Patients below 18 years old and patients above 85 years old
* Patients with type I diabetes mellitus (Insulin dependent diabetes mellitus IDDM)
* Pregnant women and lactating women diagnosed with diabetes or intending to become pregnant in the next 12 months
* Patients who had myocardial infarction within 3 months prior to screening
* Patients who had transient ischemic attack (TIA), ischemic or hemorrhagic stroke within 3 months prior to screening
* Patients with poorly controlled diabetes mellitus, defined as patients having glycosylated hemoglobin (HbA1c) level of ≥12% at screening or patients who were hospitalized for diabetic ketoacidosis or hyperosmolar coma within 4 months prior to screening
* Patients with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 at screening
* Patients with severe hepatic impairment of Child-Turcotte-Pugh class C at screening
* Patients treated with antidiabetic drugs thiazolidinediones (TZD) (rosiglitazone and pioglitazone) prior to screening
* Patients who were receiving SGLT2 inhibitors (e.g., dapagliflozin, canagliflozin, or empagliflozin) within 3 months prior to screening
* Known allergy or hypersensitivity to any component of the study drugs
* Current or previous participation in another clinical study involving the systemic or ocular administration of an investigational drug or device within 6 months of screening

Study eye exclusion criteria:

* Macular edema caused by other conditions than diabetic macular edema or coexisting with DME such as retinal vein occlusion, choroidal neovascularization (CNV), or uveitic cystoid macular edema
* History of postoperative cystoid macular edema (Irvine-Gass syndrome)
* Cataract extraction within 3 months prior to screening
* Patients who had previous macular laser treatment
* Patients who had peripheral panretinal photocoagulation laser (PRP) treatment within 6 months prior to screening
* Patients who have been treated with intravitreal anti-VEGF or intravitreal corticosteroids within 6 months prior to screening
* The use of corticosteroids or non-steroidal anti-inflammatory eye drops within 1 month prior to screening
* Patients on topical prostaglandin analogs (e.g., latanoprost, travoprost, ioprost, or tafluprost) at screening
* History of vitrectomy or scleral buckling
* Presence of diffuse vitreomacular traction or thick epiretinal membrane on OCT causing significant traction
* Presence of tractional retinal detachment involving the macula and requiring vitrectomy
* Presence of other associated macular pathology (e.g., macular scars or macular holes) on OCT
* Presence of rubeosis iridis
* Signs of hypertensive retinopathy (arterioral spasm or silver wiring of blood vessels)
* Presence of glaucoma
* Aphakia
* Yttrium aluminum garnet (YAG) laser capsulotomy within 3 months prior to screening
* Patients diagnosed with ocular surface infections until treated prior to receiving the intravitreal injections

Non-study eye exclusion criteria:

• The non-study eye receiving simultaneous intravitreal anti-VEGF treatment with the study eye

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean central subfield thickness (CST) | Baseline, 3 months
  The reduction in mean central subfield thickness (CST) from baseline will be determined using Optical Coherence Tomography (OCT) and compared between study groups.
The best-corrected visual acuity (BCVA) | Baseline, 3 months
  The improvement in the best-corrected visual acuity (BCVA) from baseline will be recorded and compared between study groups.

SECONDARY OUTCOMES:
Percentage of patients with persistent macular edema | 3 months
  The number of patients with persistent macular edema who are indicated to continue intravitreal anti-VEGF therapy beyond the initial 3 injections will be compared across study groups.
Retinal anatomical changes | Baseline, 3 months
  Retinal anatomical changes such as the improvement of cystoid macular spaces and resolution of subretinal fluid will be determined on OCT.
Visual impairment patient reported outcome | Baseline, 3 months
  Patient reported outcome measures for visual impairment will be reported at baseline and after receiving interventions, using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25), and compared across study groups.
Incidence of adverse events | 3 months
  Systemic and ocular adverse events will be recorded and compared across study groups to assess the safety profile of the interventions.
Measuring the levels of some inflammatory cytokines in the aqueous humor | Baseline, 2 months
  The routinely withdrawn aqueous humor samples from patients with DME during intravitreal anti-VEGF injection will be collected and analyzed. The levels of inflammatory cytokines VEGF-A, interleukin (IL)-6, monocyte chemoattractant protein 1 (MCP-1), and tumor necrosis factor (TNF)-α, will be quantified, using multiplex protein analysis, and compared between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Amira A. Nayel, MSc, Principal Investigator — Clinical researcher and PhD student at the Faculty of Pharmacy, Alexandria University
Locations (1):
- Alexandria Main University Hospital, The Ophthalmology Department, Faculty of Medicine, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No